CLINICAL TRIAL: NCT05413512
Title: Stressor-evoked Brain and Cardiovascular Responses to Acute Psychological Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Annie Ginty, Assistant Professor, Baylor University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1437575; K01HL145021 (NIH)
Record Dates: First submitted 2022-06-05; First posted 2022-06-10 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Acute Psychological Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute psychological stress task (MSIT; Stroop) (Experimental): Multi-source interference task (MSIT; Stroop)
  Interventions: Other: Acute psychological stress

INTERVENTIONS:
Other: Acute psychological stress — Experimental: Acute psychological stress Two, acute-psychological stress tasks known to reliably elicit a cardiovascular responses (Multi-source interference task; Stroop).

SUMMARY:
The present study will examine cardiovascular, metabolic, and neural responses to acute psychological stress using a cross-sectional approach.

DETAILED DESCRIPTION:
All participants in this study will undergo an acute psychological stress paradigm, consisting of two acute psychological stress tasks (MSIT and Stoop). There is no formal randomization since al participants are randomized to undergo the acute psychological stress tasks.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old

Exclusion Criteria:

* Chronic medical or neurological condition
* Pregnant
* Current illness or infection
* Any condition that would prohibit engaging in physical exercise
* Any metal implants in body
* Claustrophobia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Ginty, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other rsearchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited in Waco, Texas area
Pre-assignment Details: All participants engaged in the acute psychological stress task.
Groups:
- Acute Psychological Stress: Participants will undergo an acute psychological stress task that has been shown to elicit neural, cardiovascular, and psychological (feelings of stressfulness) responses.
Period: Overall Study
Arm/Group | Acute Psychological Stress
Started | 170
Completed | 170
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Acute Psychological Stress: Participants will undergo an acute psychological stress task that has been shown to elicit neural, cardiovascular, and psychological (feelings of stressfulness) responses.
  Acute psychological stress: Participants will undergo an acute psychological stress task that has been shown to elicit neural, cardiovascular, and psychological (feelings of stressfulness) responses.
Arm/Group | Acute Psychological Stress
Number analyzed (Participants) | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 170
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.08 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 132
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 103
  More than one race | 13
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 170

OUTCOME MEASURES:

1. Primary Outcome: Stressor-evoked Oxygen Consumption in mL/(kg·Min) (Stress - Baseline)
Description: Stressor-evoked oxygen consumption. (Oxygen consumption during acute psychological stress task - Oxygen consumption during resting baseline).
Time Frame: 18 minutes (approximately 9 minutes for each task)
Measure: Mean (Standard Deviation); unit: mL/(kg·min)
Groups:
- Acute Psychological Stress Task: Stressor-evoked oxygen consumption. (Oxygen consumption during acute psychological stress task - Oxygen consumption during resting baseline).
Arm/Group | Acute Psychological Stress Task
Number analyzed (Participants) | 169
mL/(kg·min)
  Stroop task | 0.265 (0.452)
  MSIT task | 0.287 (0.431)

2. Primary Outcome: Heart Rate (Bpm) Measured by Electrocardiogram
Description: Stressor-evoked heart rate. (Heart rate during acute psychological stress task - Heart rate during resting baseline).
Time Frame: 18 minutes (approximately 9 minutes for each stress task)
Population: Data loss for 3 participants due to equipment malfunction.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Acute Psychological Stress
Number analyzed (Participants) | 167
beats per minute (bpm)
  Stroop task | 4.926 (7.456)
  MSIT | 2.826 (6.317)

3. Primary Outcome: Neural Activity Measured by fMRI
Description: Stressor-evoked neural activity.
  Incongruent-vs-Congruent t at the group-level, filtered at 0.05 after FDR correction and with a cluster extent of 50 voxels.
Time Frame: 18 minutes (approximately 9 minutes for each stress task).
Population: Participants who have full data for both acute psychological stress tasks during fMRI scanning.
Measure: Mean (Standard Error); unit: BOLD signal (Incon - Con)
Arm/Group | Acute Psychological Stress
Number analyzed (Participants) | 160
BOLD signal (Incon - Con)
  L Parietal_inf (stroop) | 0.71 (0.41)
  R Angular (stroop) | 0.54 (0.35)
  R Supp_Motor_Area (stroop) | 1 (0.65)
  L Frontal_Inf_Tri (stroop) | 0.85 (0.56)
  L Parietal_Inf2 (stroop) | 0.66 (0.45)
  R Insula (stroop) | 0.70 (0.50)
  R Frontal_Inf_Oper (stroop) | 0.76 (0.60)
  R Vermis (stroop) | 0.84 (0.68)
  R Thalamus (stroop) | 0.48 (0.40)
  L Precuneus2 (stroop) | -0.55 (0.52)
  L ParaHippocampal2a (stroop) | -0.47 (0.50)
  L Angular2 (stroop) | -0.49 (0.54)
  L Frontal_Med_Orb2 (stroop) | -1.38 (1.57)
  L Frontal_Sup2 (stroop) | -0.55 (0.66)
  L ParaHippocampal2 (stroop) | -0.47 (0.58)
  R ParaHippocampal2 (stroop) | -0.35 (0.46)
  R Precentral2 (stroop) | -0.20 (0.31)
  R Rolandic_Oper2 (stroop) | -0.19 (0.33)
  R Angular2 (stroop) | -0.23 (0.45)
  R Amygdala2 (stroop) | -0.21 (0.43)
  R Frontial_Sup2 (stroop) | -0.24 (0.54)
  R Cerebelum_Crus2 (stroop) | -0.29 (0.91)
  L Parietal_Inf (MSIT) | 0.50 (0.40)
  R Parietal_Inf (MSIT) | 0.49 (0.43)
  R Angular (MSIT) | 0.35 (0.31)
  L Supp_Motor_Area (MSIT) | 0.49 (0.45)
  L Frontal_Inf_Oper (MSIT) | 0.54 (0.52)
  R Calcarine (MSIT) | 0.45 (0.48)
  R Frontal_Inf_Oper (MSIT) | 0.49 (0.53)
  R Insula (MSIT) | 0.49 (0.54)
  R Frontal_Mid (MSIT) | 0.31 (0.37)
  L Thalamus (MSIT) | 0.32 (0.39)
  L Frontal_Mid_Orb (MSIT) | 0.25 (0.53)
  L Cingulum_Mid2 (MSIT) | -0.40 (0.41)
  L Angular2 (MSIT) | -0.51 (0.62)
  L Frontal_Sup2 (MSIT) | -0.43 (0.52)
  L Frontal_Med_Orb2 (MSIT) | -1.06 (1.33)
  R Hippocampus2 (MSIT) | -0.24 (0.37)
  R Angular2 (MSIT) | -0.27 (0.46)
  R Insula2 (MSIT) | -0.21 (0.35)
  R Temporal_Mid2 (MSIT) | -0.32 (0.63)
  R Cerebellum_Crus2 (MSIT) | -0.42 (0.83)
  R Precentral2 (MSIT) | -0.10 (0.30)
  L Cerebellum_Crus2 (MSIT) | -0.26 (0.88)

ADVERSE EVENTS:
Time Frame: 4 total hours (participants were monitored during each of the 2 hour lab visits).
Arm/Group | Acute Psychological Stress
All-Cause Mortality (participants affected / at risk) | 0/170
Serious Adverse Events (participants affected / at risk) | 0/170
Other Adverse Events (participants affected / at risk) | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT05413512/Prot_SAP_000.pdf